CLINICAL TRIAL: NCT03219931
Title: Effects of an Association of the Two Bifidobacteria Probiotics Bifidobacterium Breve B632 and Bifidobacterium Breve BR03 in Intestinal Bacterial Colonization and in the Prevention and/or Reduction of the Incidence of Colics in Infants
Brief Title: NEOBIFI: Clinical Trial for the Prevention and/or Reduction of the Incidence of Colics in Infants
Acronym: NEOBIFI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Assoc. Professor in Clinical Nutrition, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE 63/13
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Colic, Infantile; Probiotic; Gut Microbiome; Bifidobacterium Breve
Keywords: infant colics; probiotic; gut microbiome; bifidobacterium breve; crying time
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: During the 90 days of the study, parents were asked to give 5 drops of active product (108 viable cells/strain) or placebo and to daily take note of minutes of crying, number, color, and consistency of evacuations, and number of regurgitations or vomits.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is a triple blind study in which the treatment or intervention is unknown to the research participant, the individuals who administer the treatment or intervention, and the researchers who assess the outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active group - Breastfeeding infants (Active Comparator): In this Group will be enrolled only infants who are breastfed. This Group will take the active product containing 5 drops of active product (108 viable cells/strain) of Bifidobacterium breve BR03 and Bifidobacterium breve B632.
  Interventions: Drug: Bifidobacterium breve BR03 and Bifidobacterium breve B632
- Active Group - Bottlefeeding infant (Active Comparator): In this active Group will be enrolled only infant who are bottle-fed. This Group will take the active product containing 5 drops of active product (108 viable cells/strain) of Bifidobacterium breve BR03 and Bifidobacterium breve B632.
  Interventions: Drug: Bifidobacterium breve BR03 and Bifidobacterium breve B632
- Placebo group - Breastfeeding infants (Placebo Comparator): In this placebo Group will be enrolled only infants who are breastfed. This arm will receive a supplementation with a same product equal to the active product but without bifidobacterium inside.
  Interventions: Drug: Placebos
- Placebo group - Bottlefeeding infants (Placebo Comparator): In this placebo Group will be enrolled only infants who are bottlefed. This arm will receive a supplementation with a same product equal to the active product but without bifidobacterium inside.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Bifidobacterium breve BR03 and Bifidobacterium breve B632 — This is the active product containing 108 viable cells/strain
  Arms: Active Group - Bottlefeeding infant; Active group - Breastfeeding infants
Drug: Placebos — This is the placebo product containing a similar product without bifidobacterium inside.
  Other Names: Placebo
  Arms: Placebo group - Bottlefeeding infants; Placebo group - Breastfeeding infants

SUMMARY:
Infant colics represent a clinical condition in childhood, characterized by an uncontrollable crying that occurs without any apparent organic cause.1 They can be associated with face redness, closed fists, thighs flexion, meteorism, and gas emission. They are generally diagnosed according to Wessel's "rule of three" (>3 h of crying a day, for >3d a week, for >3wk in a row).2 These crises tend to reach their maximum intensity at 6 weeks of age, in most cases.3 They represent a serious source of anxiety for the family, increasing hospital admissions (5.8% of infants),4 postpartum depression risk, with higher stress levels for up to 3 years from these events. The etiology is still unknown. Anyway, it's assumed that the following factors may be involved: (1) Lactose intolerance. (2) Food hypersensitivity. (3) Feeding difficulties. (4) Disorders of the enteric nervous system. (5) Alterations of pain transmission. (6) Gastroesophageal reflux. (7) Intestinal hormones. (8) Psychosocial factors. (9) Alteration of the intestinal microbiota. In 1994, Lehtonen was the first to suggest that an altered intestinal microbiota composition in the very first months may induce intestinal colics in infants. Human intestinal microbiota is composed of about 1013 to 1014 microorganisms, mainly bacteria. The total number of microbiota genes is called "microbioma" and it is estimated to be 150 times the number of genes in the human genome.5 It acts as a real organ, whose activity can be influenced by diet, lifestyle, prebiotics, probiotics, and antibiotics. Several studies revealed the predominance of bifidobacteria in breastfed infants, whereas bottle-fed infants show a mixed population where bifidobacteria are less represented. the intestinal microbiota composition in a 3-year-old child is already similar to that of an adult.6 Other factors conditioning the microbiota are gestational age and type of birth. Colicky infants have a microbiota with a slow development and a lower stability over time.7 It also contains less lactobacilli and bifidobacteria, and a prevalence of gram-negative bacteria. The stools of these children often show increased levels of calprotectin, an intestinal index of inflammation.

RISK FACTORS ARE SEVERAL: Smoking: The exposure to cigarette smoke may be related to colics; this might be connected to the increase of plasma and intestinal levels of motilin. Maternal smoking during pregnancy seems to increase the risk of developing colics, more than postnatal exposition to smoke.8

Psychosocial: Infant colics may be more frequent with an instable psychosocial family environment. Maternal stress, anxiety, and depression are important risk factors.8 Breastfeeding: The difference between breastfeeding and bottlefeeding for colicky infants is controversial. Many studies have shown contrasting results,17 but the majority of the authors agree to attribute an important role to bottlefeeding. 9 A melatonin role was assumed too. This hormone is not secreted in infants, but only in adults, and has a hypnotic and relaxing role on the gastrointestinal smooth muscle. Its concentration shows a clear circadian rhythm, with a pick during night hours. Its presence in breast milk may be related to the lower occurrence of colics in breastfed infants compared with the bottle-fed infants.9 Recent literature shows an increasing attention toward probiotics,10 for the intestinal microbiota modulation. Some Lactobacillus reuteri strains were studied, with contrasting results in different studies; other probiotics as bifidobacteria showed in vitro anti-inflammatory properties and the ability to inhibit coliforms growth, whose presence is significant in colicky infants. Some probiotics exert a direct action on the bacterial growth, through bacteriocins production and final fermentation products.11 Bifidobacterium breve was isolated from healthy infants' feces.12 Aloisio et al13 tested in vitro ability of this strain and of other 45 bifidobacteria strains to oppose the growth of several microorganisms such as E. coli, S. enteriditis, C. difficile, K. pneumoniae, and Enterobacter cloacae. B. breve BR03, in a randomized clinical study, proved to have a beneficial effect on constipation in adults, it also seemed effective for the reduction of gas formation and for abdominal distension, and no side effects were shown during the treatment, while the beneficial effects lasted for up to 15 days after the end of the treatment.14,15 Both bifidobacteria strains showed, during an in vitro study, the ability to oppose 4 strains of E. coli; in particular, BR03 displayed an activity against E. coli O157:H7, an enterohemorrhagic strain that through Shiga toxin causes a potentially lethal infection.16

DETAILED DESCRIPTION:
Type of Study: Interventional single-center, double-blind, randomized study, with treatment and placebo controlled.

Population: Only healthy babies were accepted. They were not treated with antibiotics, enrolled within 15 days from birth, and with an informed consent signed by the parents.

Parents were asked to make an initial recruitment examination within 15 days from birth and a second one at the 91st day of age, at the clinic of Pediatric Gastroenterology.

During the 90 days of the study, parents were asked to give 5 drops of active product (108 viable cells/strain) or placebo and to daily take note of minutes of crying, number, color, and consistency of evacuations, and number of regurgitations or vomits.

Probiotical S.p.A. (Novara, Italy) supplied the active product and the placebo. All data were collected in a database. Randomization was performed by an external operator of the study.

STATISTIC ANALYSIS:

Categorical variables were analyzed with the Fischer exact test. Comparisons between numeric variables between various groups were performed with the Kruskal-Wallis test (in the case of >2 groups) and with the Wilcoxon test for independent samples (in the case of only 2 groups being compared). A probability value of P<0.05 was considered as the limit of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Only healthy babies term born
* Between 6 days and 15 days of life
* With a Birth weight between 2500 gr and 4000 gr
* With natural childbirth

Exclusion Criteria:

* Adverse reactions to the product or component of the product (allergies…)
* Antibiotic treatments
* Chronic diseases, hepatic or gastroenterological diseases
* Medical treatment for chronic diseases
* Probiotic or prebiotic therapies

Ages: 6 Days to 15 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in infants crying - reduction of infants crying | Change from Baseline (V0) of infant crying at 3 months (V1)
  The primary endpoint of the study was the assessment of the effectiveness of B. breve B632 and BR03 association in the reduction of infants crying over time. Both breastfed and bottle-fed babies were studied.

SECONDARY OUTCOMES:
Change in gastrointestinal symptoms | Change from Baseline (V0) of fecal evacuations, regurgitations and vomits at 3 months (V1)
  The second endpoint was to observe the effect of these probiotics on daily evacuations and on the number of regurgitations and vomits.
Change in fecal microbiome | Change from Baseline of fecal microbiome (V0) at 3 months (V1)
  Evaluate any variation of fecal microbiome

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Maggiore della Carità - Clinica Pediatrica - Ambulatorio di Gastroenterologia Pediatrica, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savino F. Focus on infantile colic. Acta Paediatr. 2007 Sep;96(9):1259-64. doi: 10.1111/j.1651-2227.2007.00428.x. PMID 17718777
- [Background] WESSEL MA, COBB JC, JACKSON EB, HARRIS GS Jr, DETWILER AC. Paroxysmal fussing in infancy, sometimes called colic. Pediatrics. 1954 Nov;14(5):421-35. No abstract available. PMID 13214956
- [Background] Kheir AE. Infantile colic, facts and fiction. Ital J Pediatr. 2012 Jul 23;38:34. doi: 10.1186/1824-7288-38-34. PMID 22823993 (Retraction: PMID 24618350 Ital J Pediatr. 2014;40(1):9)
- [Background] Iacono G, Merolla R, D'Amico D, Bonci E, Cavataio F, Di Prima L, Scalici C, Indinnimeo L, Averna MR, Carroccio A; Paediatric Study Group on Gastrointestinal Symptoms in Infancy. Gastrointestinal symptoms in infancy: a population-based prospective study. Dig Liver Dis. 2005 Jun;37(6):432-8. doi: 10.1016/j.dld.2005.01.009. Epub 2005 Mar 2. PMID 15893282
- [Background] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603
- [Background] Brooks GF, Carroll KC, Butel JS, et al. Jawetz, Melnick, & Adelberg's Medical Microbiology, 26e. Columbus, OH: McGraw-Hill; 2013.
- [Background] de Weerth C, Fuentes S, Puylaert P, de Vos WM. Intestinal microbiota of infants with colic: development and specific signatures. Pediatrics. 2013 Feb;131(2):e550-8. doi: 10.1542/peds.2012-1449. Epub 2013 Jan 14. PMID 23319531
- [Background] Yalcin SS, Orun E, Mutlu B, Madendag Y, Sinici I, Dursun A, Ozkara HA, Ustunyurt Z, Kutluk S, Yurdakok K. Why are they having infant colic? A nested case-control study. Paediatr Perinat Epidemiol. 2010 Nov;24(6):584-96. doi: 10.1111/j.1365-3016.2010.01150.x. Epub 2010 Aug 17. PMID 20955236
- [Background] Cohen Engler A, Hadash A, Shehadeh N, Pillar G. Breastfeeding may improve nocturnal sleep and reduce infantile colic: potential role of breast milk melatonin. Eur J Pediatr. 2012 Apr;171(4):729-32. doi: 10.1007/s00431-011-1659-3. Epub 2011 Dec 29. PMID 22205210
- [Background] WHO. WHO European Ministerial Conference on Nutrition and Noncommunicable Diseases in the Context of Health 2020. Vienna: WHO; 2013.
- [Background] Sanders ME. Impact of probiotics on colonizing microbiota of the gut. J Clin Gastroenterol. 2011 Nov;45 Suppl:S115-9. doi: 10.1097/MCG.0b013e318227414a. PMID 21992949
- [Background] Scardovi V, Casalicchio F, Vincenzi N. Multiple electrophoretic forms of transaldolase and 6-phosphogluconic dehydrogenase and their relationships to the taxonomy and ecology of the bifidobacteria. Int J Syst Bacteriol. 1979;29:312-327.
- [Background] Aloisio I, Santini C, Biavati B, Dinelli G, Cencic A, Chingwaru W, Mogna L, Di Gioia D. Characterization of Bifidobacterium spp. strains for the treatment of enteric disorders in newborns. Appl Microbiol Biotechnol. 2012 Dec;96(6):1561-76. doi: 10.1007/s00253-012-4138-5. Epub 2012 May 17. PMID 22588500
- [Background] Del Piano M, Carmagnola S, Anderloni A, Andorno S, Ballare M, Balzarini M, Montino F, Orsello M, Pagliarulo M, Sartori M, Tari R, Sforza F, Capurso L. The use of probiotics in healthy volunteers with evacuation disorders and hard stools: a double-blind, randomized, placebo-controlled study. J Clin Gastroenterol. 2010 Sep;44 Suppl 1:S30-4. doi: 10.1097/MCG.0b013e3181ee31c3. PMID 20697291
- [Background] Iemoli E, Trabattoni D, Parisotto S, Borgonovo L, Toscano M, Rizzardini G, Clerici M, Ricci E, Fusi A, De Vecchi E, Piconi S, Drago L. Probiotics reduce gut microbial translocation and improve adult atopic dermatitis. J Clin Gastroenterol. 2012 Oct;46 Suppl:S33-40. doi: 10.1097/MCG.0b013e31826a8468. PMID 22955355
- [Background] Mogna L, Del Piano M, Deidda F, Nicola S, Soattini L, Debiaggi R, Sforza F, Strozzi G, Mogna G. Assessment of the in vitro inhibitory activity of specific probiotic bacteria against different Escherichia coli strains. J Clin Gastroenterol. 2012 Oct;46 Suppl:S29-32. doi: 10.1097/MCG.0b013e31826852b7. PMID 22955353
- [Background] Savino F, Cordisco L, Tarasco V, Palumeri E, Calabrese R, Oggero R, Roos S, Matteuzzi D. Lactobacillus reuteri DSM 17938 in infantile colic: a randomized, double-blind, placebo-controlled trial. Pediatrics. 2010 Sep;126(3):e526-33. doi: 10.1542/peds.2010-0433. Epub 2010 Aug 16. PMID 20713478
- [Background] Van Niel CW. Probiotics: not just for treatment anymore. Pediatrics. 2005 Jan;115(1):174-7. doi: 10.1542/peds.2004-2356. No abstract available. PMID 15629997
- [Background] Roger LC, Costabile A, Holland DT, Hoyles L, McCartney AL. Examination of faecal Bifidobacterium populations in breast- and formula-fed infants during the first 18 months of life. Microbiology (Reading). 2010 Nov;156(Pt 11):3329-3341. doi: 10.1099/mic.0.043224-0. Epub 2010 Sep 23. PMID 20864478
- [Background] Savino F, Cordisco L, Tarasco V, Calabrese R, Palumeri E, Matteuzzi D. Molecular identification of coliform bacteria from colicky breastfed infants. Acta Paediatr. 2009 Oct;98(10):1582-8. doi: 10.1111/j.1651-2227.2009.01419.x. Epub 2009 Jul 9. PMID 19604166
- [Background] Rhoads JM, Fatheree NY, Norori J, Liu Y, Lucke JF, Tyson JE, Ferris MJ. Altered fecal microflora and increased fecal calprotectin in infants with colic. J Pediatr. 2009 Dec;155(6):823-828.e1. doi: 10.1016/j.jpeds.2009.05.012. Epub 2009 Jul 22. PMID 19628216
- [Background] Indrio F, Di Mauro A, Riezzo G, Civardi E, Intini C, Corvaglia L, Ballardini E, Bisceglia M, Cinquetti M, Brazzoduro E, Del Vecchio A, Tafuri S, Francavilla R. Prophylactic use of a probiotic in the prevention of colic, regurgitation, and functional constipation: a randomized clinical trial. JAMA Pediatr. 2014 Mar;168(3):228-33. doi: 10.1001/jamapediatrics.2013.4367. PMID 24424513
- [Background] Sung V, Hiscock H, Tang ML, Mensah FK, Nation ML, Satzke C, Heine RG, Stock A, Barr RG, Wake M. Treating infant colic with the probiotic Lactobacillus reuteri: double blind, placebo controlled randomised trial. BMJ. 2014 Apr 1;348:g2107. doi: 10.1136/bmj.g2107. PMID 24690625